CLINICAL TRIAL: NCT04320992
Title: A Multicenter Prospective Study of "High Risk" Molecular Typing in Patients With Adult T Lymphoblastic Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Other Study IDs: B2020-046
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: T-Lymphoblastic Lymphoma/Leukemia
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- tested group
- controlled group

SUMMARY:
The purpose of this study is to determine the indicative value of "high risk" molecular typing in patients with adult T lymphoblastic lymphoma

ELIGIBILITY:
Inclusion Criteria:

* biopsy proved T lymphoblastic lymphoma
* newly diagnosed patients

Exclusion Criteria:

* patients with biopsy samples unavailable

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adults
Sampling Method: Probability Sample
Enrollment: 207 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 3-years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University,, Guangzhou, China